CLINICAL TRIAL: NCT04010786
Title: Investigation of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Subcutaneous Injections of NNC0247-0829 in Adults With Overweight or Obesity
Brief Title: A Research Study Investigating NNC0247-0829 for Weight Management in People With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9215-4424; U1111-1226-5167 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: First human dose trial; a single-centre, placebo-controlled, double-blind (within cohorts), randomised SD and MD ascending dose trial with a sequential trial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active treatment NNC0247-0829 (Experimental): Up to 6 single dose cohorts are planned with 10 subjects in each; 8 will receive active treatment. Up to 2 multiple dose cohorts are planned with 12 subjects in each; 8 will receive active treatment
  Interventions: Drug: NNC0247-0829
- Placebo (Placebo Comparator): In each of the 6 single dose cohorts, 2 subjects will receive placebo. In the 2 multiple dose cohorts, 4 subjects will receive placebo
  Interventions: Drug: Placebo (NNC0247-0829)

INTERVENTIONS:
Drug: NNC0247-0829 — Participants will receive either single or multiple doses given subcutaneously (s.c., under the skin) in a lifted fold of the stomach skin. Dose level and number of doses will depend on the cohort.
  Arms: Active treatment NNC0247-0829
Drug: Placebo (NNC0247-0829) — Participants will receive either single or multiple doses of placebo given s.c. in a lifted fold of the stomach skin.
  Arms: Placebo

SUMMARY:
This study looks at NNC0247-0829 (a potential new medicine) for weight management in people with overweight or obesity. The study looks at how NNC0247-0829 works in the body. Participants will either get NNC0247-0829 or placebo (a 'dummy' medicine) - which treatment is decided by chance. NNC0247-0829 is an experimental medicine which has not been approved by the US FDA. Participants will get either 1 injection or a total of 4 injections (one week apart) by a study nurse at the clinic depending on what group they are in. The study will last for about 18 months, but participation will last from 11 to 23 weeks. This will depend on the group participants are in. Participants will attend 8 to 14 visits at the clinic with the study staff. Some participants will have one 16-day, 15-night visit and one 2-day, 1-night visit. Others will have two 2-day, 1-night visits. At all visits except one, participants will have blood tests and other checks. They will be asked about their health, medical history and habits including mental health questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Female not of childbearing potential (CBP) or male, aged 18-60 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 27.0 and 34.9 kg/m^2 (both inclusive) in the SD cohorts and between 27.0 and 39.9 kg/m^2 (both inclusive) in the MD cohorts at screening. Overweight or obesity should be due to excess adipose tissue, as judged by the investigator.

Exclusion Criteria:

* Male subject who is not surgically sterilised (vasectomised) and is sexually active with female partner of childbearing potential in the absence of highly effective contraception.
* Any disorder, which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol.
* Use of prescription or non-prescription products, including herbal products and non-routine vitamins, within 14 days prior to screening. Mild painkillers are permitted until 24h prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
For single dose (SD) cohorts: Number of treatment emergent adverse events (TEAEs) | From time of first dosing (Day 1) until Day 71
  Number of events
For multiple dose (MD) cohorts: Number of treatment emergent adverse events (TEAEs) | From time of first dosing (Day 1) until Day 85
  Number of events

SECONDARY OUTCOMES:
For SD cohorts: Number of injection site reactions | From time of first dosing (Day 1) until Day 71
  Number of events
For SD cohorts: Occurrence of anti-NNC0247-0829 antibodies | From time of first dosing (Day 1) until Day 71
  Number of events
For MD cohorts: Number of injection site reactions | From time of first dosing (Day 1) until Day 85
  Number of events
For MD cohorts: Occurrence of anti-NNC0247-0829 antibodies | From time of first dosing (Day 1) until Day 85
  Number of events
For (SD) cohorts: The area under the NNC0247-0829 serum concentration-time curve from time 0 to infinity | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (from Day 71 up to Day 134, depending on the dose cohort)
  nmol/L*h

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- ICON Early Phase Services, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com